CLINICAL TRIAL: NCT02045043
Title: Genetic Risk Assessment of Defibrillator Events: A Prospective Multicenter Observational Study
Brief Title: Genetic Risk Assessment of Defibrillator Events
Acronym: GRADE
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barry London, Director, Division of Cardiovascular Medicine, University of Iowa
Other Study IDs: GRADE; R01HL077398 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Sudden Cardiac Death; Arrhythmias; Congestive Heart Failure; Cardiomyopathy
Keywords: Sudden Cardiac Death; Arrhythmias; Congestive Heart Failure; Cardiomyopathy; Single Nucleotide Polymorphisms; Genomics
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmias, Cardiac; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood was obtained for DNA (all subjects) and serum (subgroup of subjects)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiomyopathy patients with ICDs

SUMMARY:
Arrhythmias remain a major health problem, causing at least 250,000 deaths annually in the United States. Pharmacological treatments often do more harm than good, and device therapies are limited by high cost and effects on quality of life. Ion channel mutations cause rare inherited arrhythmopathies, but account for only a small fraction of patients with life- threatening arrhythmias and sudden death. Most arrhythmias occur during myocardial ischemia, following myocardial infarction, and in patients with poor left ventricular (LV) function of any etiology. Aside from ejection fraction (EF), few clinically useful indicators to stratify the risk of sudden death have been identified. The role of subtle difference in ion channel expression and/or structure in predisposing patients to arrhythmias and modulating the risk of sudden death is unknown.

In this study, we are prospectively testing whether polymorphisms in ion channels and ion channel modifying genes are associated with arrhythmias in a population with internal cardioverter-defibrillators (ICDs) and poor LV function. We will test the hypothesis that functional polymorphisms in the coding sequences and promoter regions of cardiac genes (e.g. ion channels, beta-adrenergic receptors) predispose individuals to arrhythmias and /or heart failure progression.

We hope to identify genetic predictors for the common forms of sudden cardiac death. This would allow the identification of a subpopulation of heart failure patients that would benefit most from ICD placement.

ELIGIBILITY:
Inclusion Criteria:

* An ICD placed during the last 5 years, or a planned ICD within 1 month
* Age 18 or older
* Left Ventricular Ejection fraction < or = 30%
* Ability to give informed consent

Exclusion Criteria:

* Patient refuses or is unable to give consent
* A life expectancy <6 months from a non-cardiac life threatening disease
* Ongoing Class IV heart failure symptoms despite treatment
* History of cardiac transplant or left ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age and over with a cardiomyopathy, an ejection fraction less than or equal to 30%, and an implantable cardioverter defibrillator
Sampling Method: Non-Probability Sample
Enrollment: 1807 (Actual)
Dates: Start 2002-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Shock-Free Survival | Up to 5 years
  Time to first appropriate shock from an Implantable Cardioverter-Defibrillator

SECONDARY OUTCOMES:
Survival | Up to 5 years
  Time to death from any cause
Transplant- and VAD-Free Survival | Up to 5 years
  Time to occurence of death from any cause, cardiac transplantation, or Ventricular Assist Device placement (whichever comes first)
Appropriate Shock Frequency | Up to 5 years
  The number of appropriate shocks per year

CONTACTS AND LOCATIONS:
Overall Officials: Barry London, MD PhD, Principal Investigator — University of Iowa
Locations (6):
- United States (6):
  - Emory University, Atlanta, Georgia
  - Massuchetts General Hospital, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
  - Mid Ohio Cardiology, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Refaat MM, Lubitz SA, Makino S, Islam Z, Frangiskakis JM, Mehdi H, Gutmann R, Zhang ML, Bloom HL, MacRae CA, Dudley SC, Shalaby AA, Weiss R, McNamara DM, London B, Ellinor PT. Genetic variation in the alternative splicing regulator RBM20 is associated with dilated cardiomyopathy. Heart Rhythm. 2012 Mar;9(3):390-6. doi: 10.1016/j.hrthm.2011.10.016. Epub 2011 Oct 17. PMID 22004663
- [Result] Blanco RR, Austin H, Vest RN 3rd, Valadri R, Li W, Lassegue B, Song Q, London B, Dudley SC, Bloom HL, Searles CD, Zafari AM. Angiotensin receptor type 1 single nucleotide polymorphism 1166A/C is associated with malignant arrhythmias and altered circulating miR-155 levels in patients with chronic heart failure. J Card Fail. 2012 Sep;18(9):717-23. doi: 10.1016/j.cardfail.2012.06.531. Epub 2012 Aug 9. PMID 22939041
- [Result] Bloom HL, Shukrullah I, Veledar E, Gutmann R, London B, Dudley SC. Statins Decrease Oxidative Stress and ICD Therapies. Cardiol Res Pract. 2010;2010:253803. doi: 10.4061/2010/253803. Epub 2010 Mar 25. PMID 20369058
- [Derived] Aleong RG, Mulvahill MJ, Halder I, Carlson NE, Singh M, Bloom HL, Dudley SC, Ellinor PT, Shalaby A, Weiss R, Gutmann R, Sauer WH, Narayanan K, Chugh SS, Saba S, London B. Left Ventricular Dilatation Increases the Risk of Ventricular Arrhythmias in Patients With Reduced Systolic Function. J Am Heart Assoc. 2015 Jul 31;4(8):e001566. doi: 10.1161/JAHA.114.001566. PMID 26231842
- [Derived] AlJaroudi WA, Refaat MM, Habib RH, Al-Shaar L, Singh M, Gutmann R, Bloom HL, Dudley SC, Ellinor PT, Saba SF, Shalaby AA, Weiss R, McNamara DM, Halder I, London B; Genetic Risk Assessment of Defibrillator Events Investigators. Effect of angiotensin-converting enzyme inhibitors and receptor blockers on appropriate implantable cardiac defibrillator shock in patients with severe systolic heart failure (from the GRADE Multicenter Study). Am J Cardiol. 2015 Apr 1;115(7):924-31. doi: 10.1016/j.amjcard.2015.01.020. Epub 2015 Jan 15. PMID 25682436